CLINICAL TRIAL: NCT05111561
Title: A Phase 1 Study of ZEN003694 in Combination With Binimetinib in Solid Tumors With RAS Pathway Alterations and Triple Negative Breast Cancer
Brief Title: Testing the Combination of the Anticancer Drugs ZEN003694 and Binimetinib in Patients With Advanced/Metastatic or Unresectable Solid Tumors With RAS Alterations and Triple Negative Breast Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Amendment needed to add new dose level.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-11793; NCI-2021-11793 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10449 (Other: University of Texas MD Anderson Cancer Center LAO); 10449 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-11-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Triple-Negative Breast Carcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — binimetinib; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ZEN-3694, binimetinib) (Experimental): Patients receive ZEN-3694 PO QD and binimetinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. During the dose expansion phase, patients will have two mandatory biopsies - one before beginning the study and the second at day 15 of cycle 1. The study biopsy takes small pieces of cancer tissue from patient's body to look for markers (substances made by, on, or in tumor cells) related to how the study treatment works. Patients also undergo collection of blood samples at screening and on study and undergo CT or MRI throughout the trial.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of ZEN003694 in combination with binimetinib in treating patients with solid tumors that carry RAS alterations and that have spread to other places in the body (advanced/metastatic) or cannot be removed by surgery (unresectable). ZEN003694 is an oral medication with potential anticancer activity. It is an inhibitor of a family of proteins called bromodomain and extra-terminal (BET) which play important role during development and cellular growth. ZEN003694 may stop the growth of tumor cells that produce BET. Binimetinib is in a class of medications called kinase inhibitors. It works by blocking the action proteins called MEK1 and MEK2, that signal cancer cells to multiply. It may help keep cancer cells from growing and spreading. There is pre-clinical evidence that using ZEN003694 and binimetinib together may shrink or stabilize cancers studied in this trial. There are two parts of this study; dose escalation and dose expansion. In the dose escalation part of this study, different people will get different doses of the study drugs ZEN003694 and binimetinib. In the dose expansion part of this study, the highest dose with manageable side effects will be given to additional people. This will help to understand the side effects that may happen with this drug combination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of BET bromodomain inhibitor ZEN-3694 (ZEN003694 [ZEN-3694]) and binimetinib when given in combination in patients with advanced or metastatic solid tumors with rat sarcoma virus oncogene homolog (RAS) pathway alterations. (Part 1 [Dose Escalation]) II. To evaluate the safety and toxicity of ZEN003694 (ZEN-3694) and binimetinib when given in combination. (Part 2 [Dose Expansion])

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of ZEN003694 (ZEN-3694) and binimetinib when given in combination in patients with advanced or metastatic solid tumors with RAS pathway alterations. (Part 1 [Dose Escalation]) II. To characterize the pharmacokinetics (PK) of ZEN003694 (ZEN-3694) when given in combination with binimetinib. (Part 1 [Dose Escalation]) III. To observe and record the preliminary antitumor activity of ZEN003694 (ZEN-3694) and binimetinib when given in combination. (Part 1 [Dose Escalation]) IV. To determine the effects of ZEN003694 (ZEN-3694) and binimetinib when given in combination on patient survival and other metrics of clinical activity. (Part 2 [Dose Expansion]) IVa. To evaluate objective response rate (ORR); IVb. To evaluate progression-free survival (PFS); IVc. To evaluate duration of response (DOR); IVd. To evaluate disease control rate (DCR) at 4 months.

EXPLORATORY OBJECTIVES:

I. To characterize the PK of the ZEN003694 (ZEN-3694) and binimetinib combination. (Part 2 [Dose Expansion]) II. To identify biomarkers of sensitivity and response to the ZEN003694 (ZEN-3694) and binimetinib combination. (Part 2 [Dose Expansion]) III. To determine histone H3 acetylated at lysine 27 (H3K27ac) levels via chromatin immunoprecipitation sequencing (ChIPseq) on tumor biopsy specimen. (Part 2 [Dose Expansion]) IV. To determine the open chromatin regions in response to the ZEN003694 (ZEN-3694) and binimetinib combination using assay for transposase-accessible chromatin sequencing (ATACseq). (Part 2 [Dose Expansion])

OUTLINE: This is a dose-escalation study of ZEN-3694 with fixed dose binimetinib followed by a dose expansion.

Patients receive ZEN-3694 orally (PO) once daily (QD) and binimetinib PO twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. During the dose expansion phase, patients will have two mandatory biopsies - one before beginning the study and the second at day 15 of cycle 1. The study biopsy takes small pieces of cancer tissue from patient's body to look for markers (substances made by, on, or in tumor cells) related to how the study treatment works. Patients also undergo collection of blood samples at screening and on study and undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced/metastatic or unresectable solid tumor that is refractory to standard therapy or has relapsed after standard therapy
* Patients must have one of the following:

  * For Part 1 and 2 -

    * Triple negative breast cancer (TNBC) (estrogen receptor =< 1%, progesterone receptor =< 1%, human epidermal growth factor receptor 2 0-1+ or non-amplified)
    * Solid tumor with genomic alteration(s) activating RAS signaling including activating KRAS, NRAS, HRAS, or BRAF mutations, inactivating NF1 mutations, or BRAF fusions

      * Genomic alterations should be identified locally by next generation sequencing (NGS). Patient genomic reports will be reviewed by the MD Anderson Cancer Center (MDACC) Precision Oncology Decision Support team prior to initiation of study treatment
* For Part 1, patients can have evaluable or measurable disease. For Part 2, patients must have measurable disease by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Patients must be >= 4 weeks beyond treatment with any chemotherapy (6 weeks for nitrosoureas or mitomycin C) or other investigational therapy to include hormonal, biological, or targeted agents; or at least 5 half-lives from hormonal, biological, or targeted agents, whichever is shorter at the time of study treatment initiation. Patients must be >= 4 weeks beyond radiotherapy
* Age >= 18 years. Because no dosing or adverse events (AE) data are currently available on the use of binimetinib and ZEN003694 (ZEN-3694) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 125,000/mcL
* Hemoglobin >= 8 g/dL or >= 5.6 mmol/L
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) OR < 2.0 x ULN in patients with documented Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Calculated creatinine clearance >= 60 mL/min/1.73 m^2 (based on the calculated Chronic Kidney Disease-Epidemiology collaboration [CKD-EPI] glomerular filtration rate estimation)
* Prothrombin time =< 1.5 x ULN
* Partial thromboplastin time =< 1.5 x ULN
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this study
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to the first dose of study treatment. This exception does not include carcinomatous meningitis and primary CNS cancers, which are excluded regardless of clinical stability
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this study
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Patients must have corrected QT (QTcF) < 450 msec
* The effects of ZEN003694 (ZEN-3694) and binimetinib on the developing human fetus are unknown. For this reason and because BETi agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after the completion of ZEN003694 (ZEN-3694) and binimetinib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ZEN003694 (ZEN-3694) and binimetinib administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have not recovered from adverse events (AEs) due to prior anticancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia and peripheral neuropathy
* Patients who are receiving any other investigational agents
* Breast cancer patients with a prior history of hormone receptor positivity will not be eligible
* Patients with known PI3K pathway activating genomic alterations including inactivating mutations/deletions in PTEN and PIK3R1, amplifications in PIK3CA, and activating mutations in PIK3CA, Akt, or mTOR will not be eligible
* Prior therapy with BET, RAF, MEK, or ERK inhibitor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 (ZEN-3694) and binimetinib
* Patients requiring therapeutic doses of anticoagulation are excluded. Patients taking low-dose (prophylactic) anticoagulation (e.g., low-molecular weight heparin, low-dose warfarin, fondaparinux) are allowed. Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers). As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Patients should avoid medications that prolong the QT
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because ZEN003694 (ZEN-3694) and binimetinib are a BETi and MEK inhibitor agent, respectively, with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with ZEN003694 (ZEN-3694) and binimetinib, breastfeeding should be discontinued if the mother is treated with ZEN003694 (ZEN-3694) and binimetinib
* Patient has a history of cerebrovascular accident, myocardial infarction, or unstable angina within the previous 6 months prior to study treatment initiation
* Patients with any medical condition or diagnosis that would likely impair absorption of an orally administered drug (e.g., gastrectomy, ileal bypass, chronic diarrhea, gastroparesis) are excluded
* Patient has a history of retinal vein occlusion
* Patient has a history of pneumonitis or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (Part 1 [Dose Escalation]) | Up to 28 days from treatment start date
  Defined as the incidence of clinically significant adverse events or abnormal laboratory values thought to be at least possibly related to the study treatment occurring during the first cycle.
Incidence of adverse events (Part 2 [Dose Expansion]) | Up to 30 days after last treatment dose
  Including but not limited to treatment-emergent AEs, severe adverse events (SAEs), deaths, and clinical laboratory abnormalities, as assessed by the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) (Part 1 [Dose Escalation]) | Up to 30 days after last treatment dose
  Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Toxicity will be summarized by grade and type using descriptive statistics, including frequency and 95% confidence interval.
Pharmacokinetic (PK) parameters (Part 1 [Dose Escalation]) | Days 2, 8, 15, and 16 of cycle 1
  PK parameters will be estimated using non-compartmental method(s) and correlated with PD endpoints using non-parametric statistics.
Overall response rate (ORR) | Up to 2 years from treatment start date
  Defined as the percentage of participants who have a partial or complete response to the treatment. Descriptive statistics will be used to summarize ORR.
Disease control rate (DCR) | Up to 4 months from treatment start date
  Defined as the percentage of participants that have achieved complete response, partial response or stable disease after treatment. Descriptive statistics will be used to summarize DCR.
Duration of response (DOR) | Up to 2 years from treatment start date
  Defined as the length of time from treatment start date during the which the tumor does not grow. Kaplan-Meier method will be used to estimate DOR.
Progression free survival (PFS) | Up to 2 years from treatment start date
  Defined as the length of time during and after the study treatment during which the tumor does not grow. Kaplan-Meier method will be used to estimate PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (4):
- United States (4):
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm